CLINICAL TRIAL: NCT04106089
Title: Sleep in Pediatric Hematopoietic Stem Cell Transplant Patients
Brief Title: Sleep in Pediatric HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Rutgers University (Other); NJ Dept of Health Commission on Cancer Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-015878; DCHS20PPR006 (Other Grant/Funding Number: NJ Dept of Health Commission on Cancer Research)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Sleep; Stem Cell Transplant Complications

STUDY DESIGN:
Intervention Model Description: Aggregated N of 1 design (ABA or AAB)
Who Masked: Outcomes Assessor
Masking Description: actigraphy scoring will be conducted by study staff blind to patient study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation-Intervention-Observation (Experimental): 5 days of observation, 5 days of extended vitals check, 5 days returning to regular vitals checks
  Interventions: Behavioral: Extended time between vitals check
- Observation-Observation-Intervention (Experimental): 5 days of observation, 5 more days of observation, 5 days of extended vitals check
  Interventions: Behavioral: Extended time between vitals check

INTERVENTIONS:
Behavioral: Extended time between vitals check — Participants will have 6 hours protected sleep time (vitals checks moved from every 4 to every 6 hours)

SUMMARY:
Through an aggregated N=1 randomized controlled design (each patient will serve as their own control, with the 5-day intervention period determined by randomization), the current study will test the acceptability, feasibility, and impact on sleep and supportive care engagement of protecting one 6-hour window for nighttime sleep (intervention) relative to regular vitals checks (observation only periods) during Hematopoietic Stem Cell Transplant (HSCT) recovery.

DETAILED DESCRIPTION:
Context: Patients undergoing treatment for cancer face disease, treatment, and environmental obstacles to sufficient, sound sleep. Hospitalizations can further worsen sleep quality and quantity due to overnight vitals checks, medication administration, blood draws, and environmental noise and light. For patients undergoing hematopoietic stem cell transplant (HSCT), the risk for poor sleep is especially high due to protracted hospitalization, frequent vitals checks resulting in multiple night awakenings, and high symptom burden peaking approximately 10 days post-transplant.

Objectives:

Primary: Test the acceptability and feasibility of protecting one 6-hour window for nighttime sleep (intervention) relative to regular vitals checks (observation only periods) during HSCT recovery.

Secondary: Assess the effect of one 6-hour window for nighttime sleep on subject sleep and engagement in supportive care on the oncology unit.

Study Design:

Aggregated N=1 randomized controlled design. All participants will undergo a 5 day observation and then be randomized to receive the 5 day intervention (extended vitals checks) during either nights of days +5-+9 or days +10-+14.

Setting/Participants:

Inpatients on the HSCT Unit at the Children's Hospital of Philadelphia (CHOP)

Study Interventions and Measures:

Intervention-increasing time between vitals checks from every 4 hours to one 6-hour period at night.

Subjects will wear an actigraph for the duration of the study, complete a daily sleep diary, and complete self- and parent-proxy psychosocial measures (symptom burden, health related quality of life, sleep) and acceptability. Medical record review will also be conducted to assess vitals check frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 8 to 21 years.
2. Undergoing HSCT at The Children's Hospital of Philadelphia
3. Parent/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. History of developmental delays given the relationship to sleep/wake patterns
2. Sleep disorder diagnosis as documented in the medical record
3. Cognitive delays that impact the ability to complete study measures
4. Not proficient in English

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Barakat, PhD, Principal Investigator — CHOP
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daniel LC, Venella KL, Woodard K, Poliakova P, Gross JY, Bercovitz IN, Moore D, Barakat LP, Freedman JL. Can extending time between vital sign checks improve sleep in hematopoietic stem cell transplant patients? Testing feasibility, acceptability, and preliminary efficacy. Pediatr Blood Cancer. 2024 Apr;71(4):e30832. doi: 10.1002/pbc.30832. Epub 2024 Jan 10. PMID 38197636

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Started | 29 | 21
Completed | 21 | 19
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention | Total
Number analyzed (Participants) | 29 | 21 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.38 (3.50) | 13.62 (3.69) | 14.06 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 18 | 8 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 13 | 25
  Black | 10 | 5 | 15
  Asian | 4 | 3 | 7
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 21 | 50

OUTCOME MEASURES:

1. Primary Outcome: Patient Acceptability Questionnaire
Description: Brief questionnaire created for this study evaluating the patient's acceptability of adjusting vitals checks. Participants reported agreement with each statement on a 5-point likert scale from not at all (1) to extremely (5). Higher values indicate greater agreement.
Time Frame: 15 days after transplant
Population: 40 patients completed the full study and reported on acceptability at day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 22 | 18
units on a scale | 3.63 (1.61) | 3.55 (1.46)

2. Primary Outcome: Parent Acceptability Questionnaire
Description: as for outcome 1
Time Frame: 15 days after transplant
Population: 40 patients completed the study, but not all patients had a parent participate, thus the total number of parents reporting data is 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 19 | 18
units on a scale | 4.15 (0.89) | 3.88 (1.23)

3. Primary Outcome: Nurse Acceptability Questionnaire
Description: Brief questionnaire created for this study evaluating the nurse's acceptability of adjusting vitals checks. Nurses reported agreement with each statement on a 5-point likert scale from not at all (1) to extremely (5). Higher values indicate greater agreement.
Time Frame: 15 days after transplant
Population: 40 patients completed the full study, this is data reported by nurses about those 40 patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 22 | 18
units on a scale | 3.89 (0.96) | 3.98 (0.90)

4. Primary Outcome: Health-related Quality of Life (HRQL)
Description: Using the Pediatric Quality of Life Inventory - Stem Cell Transplant (SCT) module. Scale values range from 0 to 100, with higher scores indicating better functioning.
Time Frame: 15 days after transplant
Population: 40 participants who completed the study completed this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 22 | 18
units on a scale | 76.22 (17.13) | 72.02 (13.48)

5. Secondary Outcome: Actigraphy Sleep Efficiency
Description: Sleep efficiency is the percentage of time spent asleep, while in bed. It is calculated by dividing the time spent asleep, by the total amount of time in bed.
Time Frame: Day of the transplant through 15 days after the transplant
Population: 27 of 40 patients who completed the study had evaluable actigraphy data, presented here
Measure: Mean (Standard Deviation); unit: percentage of time in bed spent asleep
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 10 | 17
percentage of time in bed spent asleep | 74.63 (19.02) | 80.56 (16.64)

6. Secondary Outcome: Actigraphy Total Sleep Time
Description: This will measure the total amount of time the subject sleeps each day in minutes.
Time Frame: Day of the transplant through 15 days after the transplant
Population: 27 of 40 patients who completed the study had evaluable actigraphy data, presented here
Measure: Mean (Standard Deviation); unit: minutes slept per day
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 10 | 17
minutes slept per day | 374.43 (150.31) | 474.19 (141.11)

7. Secondary Outcome: Actigraphy Awakenings-minutes Per Day
Description: This measure the number of minutes per day the subject awakens from rest during nighttime sleep per day.
Time Frame: Day of the transplant through 15 days after the transplant
Population: 27 of 40 patients who completed the study had evaluable actigraphy data, presented here
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
Number analyzed (Participants) | 10 | 17
minutes per day | 122.44 (100.21) | 108.94 (96.66)

ADVERSE EVENTS:
Time Frame: During the 15 day study period.
Arm/Group | Observation-Intervention-Observation | Observation-Observation-Intervention
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/21
Other Adverse Events (participants affected / at risk) | 0/29 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04106089/Prot_SAP_000.pdf